CLINICAL TRIAL: NCT07399405
Title: Comparison of Nutrient Content Between Preterm and Term Human Milk: a Systematic Review and Meta-analysis
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Cai, Principal Investigator, Sun Yat-sen University
Other Study IDs: HMP
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Comparative Nutrient Composition of Preterm and Term Human Milk
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lactating mothers or mothers providing human milk
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — This study is a systematic review and meta-analysis. No intervention is administered to participants. Data regarding human milk composition are extracted and synthesized from previously published observational studies.

SUMMARY:
The purpose of this study is to thoroughly evaluate nutrient disparities between preterm and term human milk.

DETAILED DESCRIPTION:
Preterm birth (gestational age of less than 37 weeks) is a major global health issue, associated with a high burden of mortality and long-term morbidity. Achieving optimal nutrition is critical for improving outcomes in this vulnerable population. However, the specific nutritional requirements for supporting postnatal growth akin to intrauterine rates are exceptionally high. While human milk is the recommended foundation of nutrition, its unfortified use may not meet these demands, and common alternatives like preterm formula present a balance of potential benefits and risks. Crucially, formulating effective nutritional strategies hinges on a precise understanding of the composition of preterm human milk itself. Existing evidence on this composition, especially regarding micronutrients and their influencing factors, is inconsistent and incomplete. Prior reviews have largely focused on macronutrients, leaving a gap in the synthesized evidence regarding micronutrient levels and their key determinants. Therefore, we performed this systematic review and meta-analysis to quantitatively compare the nutrient profile of preterm and term human milk and to evaluate the influence of factors such as lactation stage on these differences.

ELIGIBILITY:
Inclusion Criteria:

* Studies needed to be population-based observational designs and report nutrient composition data for both preterm and term human milk. They must clearly define gestational age (preterm: 25-36 weeks; term: 37-42 weeks) and examine at least one comparable nutrient in both groups, such as energy, macronutrients (such as protein, fat, lactose), and/or micronutrients (including minerals like calcium and phosphorus, and vitamins such as vitamin D). We included articles published in Chinese or English only.

Exclusion Criteria:

* Studies were excluded if they focused solely on mothers with specific medical conditions (such as malnutrition, mastitis, or diabetes), if they involved nutrient supplementation as an intervention, or if they were published in languages other than Chinese or English.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Eligibility for this meta-analysis is based on the physiological capacity to produce human milk following childbirth. Therefore, the study population is inherently limited to individuals who have given birth and are lactating. This criterion is defined by biological sex (female) and obstetric history, not by gender identity. We acknowledge that this excludes individuals whose gender identity may not align with this biological capability.
Study Population: Among these studies, most of them were performed in Europe. The sample size ranged from 10 to 2,633, with a median sample size of 49. All studies provided comparative data from mothers who delivered preterm and term infants, with gestational age consistently categorized as preterm (<37 weeks) and term (≥37 weeks). The stage of lactation at sample collection (including colostrum, transitional, and mature milk) was reported in most studies.
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Energy content in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The energy content in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Protein in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of protein in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Fat in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of fat in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Lactose in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of lactose in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.

SECONDARY OUTCOMES:
Concentration of IgA in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of IgA in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Total nitrogen in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of total nitrogen in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Lysozyme in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of lysozyme in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Lactoferrin in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of lactoferrin in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Lactalbumin in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of lactalbumin in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Albumin in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of albumin in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Sodium in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of sodium in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Potassium in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of potassium in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Calcium in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of calcium in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Magnesium in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of magnesium in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Phosphorus in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of phosphorus in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Zinc in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of zinc in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Copper in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of copper in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Iron in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of iron in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Iodine in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of iodine in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Selenium in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of selenium in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Manganese in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of manganese in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Molybdenum in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of molybdenum in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Vitamin E in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of vitamin E in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Vitamin A in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of vitamin A in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.
Concentration of Vitamin B6 in human milk | Human milk samples are collected during the defined lactation periods. Specifically, colostrum is defined as samples collected within 3-5 days postpartum, transitional milk within 7-14 days postpartum, and mature milk at ≥15 days postpartum.
  The concentration of vitamin B6 in human milk. Data will be extracted from included observational studies and expressed as mean ± standard deviation for comparison between preterm and term groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No